CLINICAL TRIAL: NCT00428974
Title: A Phase 2, Randomized, Double-Blind, Dose-Ranging, Placebo-Controlled Study of the Safety and Activity of Daily CF101 Administered Orally in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: Safety and Efficacy Study of CF101 to Treat Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-201PS
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CF101 1 mg (Experimental)
  Interventions: Drug: CF101 1mg
- CF101 2mg (Experimental)
  Interventions: Drug: CF101 2mg
- CF101 4mg (Experimental)
  Interventions: Drug: CF101 4mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 1mg — CF101 1 mg q12 hours for 12 weeks
  Other Names: IB-MECA
  Arms: CF101 1 mg
Drug: CF101 2mg — CF101 2 mg q12 hours for 12 weeks
  Other Names: IB-MECA
  Arms: CF101 2mg
Drug: CF101 4mg — CF101 4 mg q12 hours for 12 weeks
  Other Names: IB-MECA
  Arms: CF101 4mg
Drug: Placebo — Placebo tablets q12 hours for 12 weeks
  Other Names: Inactive pill
  Arms: Placebo

SUMMARY:
This study will test the hypothesis that CF101, which is under development to treat other immune-mediated inflammatory diseases, will provide clinical benefits in the treatment of chronic plaque psoriasis. Patients with psoriasis who qualify for the study will be treated every 12 hours (q12h) with CF101 capsules, or placebo capsules, for 12 weeks. The safety of treatment will be carefully assessed through clinical and laboratory monitoring. The effect of treatment on psoriasis will be evaluated through standard techniques of examination and measurement of the severity of skin involvement.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, dose-ranging, placebo-controlled, study in adult males and females, ages 18 to 70 years, inclusive, with a diagnosis of moderate-to-severe chronic plaque psoriasis. At the Screening Visit, patients who provide written informed consent will have screening procedures performed, including a complete medical history, medication history, physical examination, including height, weight, blood pressure, pulse rate and temperature, and clinical laboratory tests.

Eligible patients will be those who have not received systemic retinoids, corticosteroids, or immunosuppressants (e.g., methotrexate, cyclosporine) within 6 weeks prior to initiation of study; or high potency topical corticosteroids (Class I-III), keratolytics, or coal tar (other than on the scalp, palms, groin, and/or soles); and UV or Dead Sea therapy within 4 weeks prior to initiation of study treatment. Eligible patients will be sequentially assigned to 1 of 3 dosing cohorts:

Cohort 1: CF101 1 mg (15 patients) or Placebo (5 patients); Cohort 2: CF101 2 mg (15 patients) or Placebo (5 patients); Cohort 3: CF101 4 mg (15 patients) or Placebo (5 patients).

Medication will be taken orally q12h for 12 weeks. Disease activity will be assessed using the Psoriasis Area and Severity Index (PASI) and the Physician Global Assessment (PGA). Patients will return for assessments at Weeks 2, 4, 8, 12 and 14.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 70 years of age, inclusive;
* Diagnosis of moderate-to-severe chronic plaque-type psoriasis with body surface area involvement ≥10%, as judged by the Investigator;
* Duration of psoriasis of at least 6 months;
* PASI score ≥10;
* Body weight ≤100 kg;
* Candidate for systemic treatment or phototherapy for psoriasis;
* ECG is normal or shows abnormalities which, in the judgment of the Investigator, are not clinically significant;
* Females of child-bearing potential must have a negative serum pregnancy test at screening;
* Females of child-bearing potential must be willing to use 2 methods of contraception deemed adequate by the Investigator (for example oral contraceptive pills plus a barrier method) to be eligible for, and continue participation in, the study;
* Ability to complete the study in compliance with the protocol; and
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Erythrodermic, guttate, palmar, plantar, or generalized pustular psoriasis;
* Treatment with systemic retinoids, corticosteroids, or immunosuppressants (e.g., methotrexate, cyclosporine) within 6 weeks of the Baseline visit;
* Treatment with high potency topical corticosteroids (Class I-III), keratolytics, or coal tar (other than on the scalp, palms, groin, and/or soles) within 2 weeks of the Baseline visit;
* Ultraviolet or Dead Sea therapy within 4 weeks of the Baseline visit, or anticipated need for either of these therapies during the study period;
* Treatment with a biological agent (including etanercept, adalimumab, efalizumab, infliximab, or alefacept) within a period of time equal to 5 times its circulating half-life, or 30 days, whichever is longer, prior to the Baseline visit;
* History of poor clinical response to methotrexate after an adequate regimen and duration of treatment;
* Treatment with systemic nonsteroidal anti-inflammatory drugs, beta-blockers, lithium, hydroxychloroquine, chloroquine, or systemic terbinafine within 2 weeks of the Baseline visit, or anticipated need for such drugs during the study period;
* Presence or history of uncontrolled asthma;
* Presence or history of uncontrolled arterial hypertension or symptomatic hypotension;
* Significant cardiac arrhythmia or conduction block, congestive heart failure (New York Heart Association Class 3-4), or any other evidence of clinically significant heart disease or clinically significant findings on screening electrocardiogram;
* Hemoglobin level <9.0 gm/L;
* Platelet count <125,000/mm^3;
* White blood cell count <3500/mm^3;
* Serum creatinine level greater than 1.5 times the laboratory's upper limit of normal;
* Liver aminotransferase levels greater than 2 times the laboratory's upper limit of normal;
* Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the Investigator;
* History of malignancy within the past 5 years (excluding basal cell carcinoma of the skin and ≤3 cutaneous squamous cell carcinomas, all of which have been completely excised);
* Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise patient safety, limit the patient's ability to complete the study, and/or compromise the objectives of the study;
* Participation in another investigational drug or vaccine trial concurrently or within 30 days; or within 5 half lives of a biological investigational product, whichever is longer;
* Other conditions which would confound the study evaluations or endanger the safety of the patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael David, MD, Principal Investigator — Rabin Medical Center
Locations (4):
- Israel (4):
  - Haemek Medical Center, Afula
  - Wolfson Medical Center, Holon
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Result] David M, Akerman L, Ziv M, Kadurina M, Gospodinov D, Pavlotsky F, Yankova R, Kouzeva V, Ramon M, Silverman MH, Fishman P. Treatment of plaque-type psoriasis with oral CF101: data from an exploratory randomized phase 2 clinical trial. J Eur Acad Dermatol Venereol. 2012 Mar;26(3):361-7. doi: 10.1111/j.1468-3083.2011.04078.x. Epub 2011 Apr 20. PMID 21504485

RESULTS

PARTICIPANT FLOW:
Groups:
- CF101 1 mg Twice Daily (BID); CF101 2 mg BID; CF101 4 mg BID; Placebo: Oral tablets given every 12 hours for 12 weeks
Period: Overall Study
Arm/Group | CF101 1 mg Twice Daily (BID) | CF101 2 mg BID | CF101 4 mg BID | Placebo
Started | 25 (one patient was randomized but never received study treatment) | 17 | 15 | 19
Completed | 17 | 17 | 14 | 16
Not Completed | 8 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF101 1 mg Twice Daily (BID) | CF101 2 mg BID | CF101 4 mg BID | Placebo | Total
Number analyzed (Participants) | 24 | 17 | 15 | 19 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 14 | 17 | 66
  >=65 years | 5 | 1 | 1 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (12.0) | 48.4 (10.2) | 45.3 (12.1) | 51.2 (10.4) | 49.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 5 | 5 | 17
  Male | 19 | 15 | 10 | 14 | 58
Region of Enrollment [Number; unit: participants]
  Israel | 24 | 17 | 15 | 19 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) in Psoriasis Area and Severity Index (PASI) Score
Description: PASI scale is sum of redness, thickness, and scale scores, ranging from 0 (no disease) to 72 (most severe possible score); lower scores, i..e., negative change from baseline, indicate improvement
Time Frame: 12 weeks minus baseline
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | CF101 1 mg Twice Daily (BID) | CF101 2 mg BID | CF101 4 mg BID | Placebo
Number analyzed (Participants) | 24 | 17 | 15 | 19
Scores on a scale | -0.67 (8.9) | -8.8 (7.0) | -4.1 (7.8) | -2.7 (9.4)
Statistical Analysis 1: Comparison: CF101 2 mg BID vs Placebo; 12 weeks, 2mg CF101 vs. Placebo; Test type: Superiority; p = 0.031, t-test, 1 sided

2. Secondary Outcome: The Number of Patients Who Achieve a Score of "Almost Clear" or "Clear" by Physician's Global Assessment (PGA)
Description: PGA is a scale from 0 (clear, no disease) to 5 (most severe score); patients who improve to 0 (clear) or 1 (minimal disease) are tabulated in this outcome
Time Frame: 12 weeks
Measure: Number; unit: Number of treated patients
Groups:
- CF101 1 mg BID; CF101 2 mg BID; CF101 4 mg BID; Placebo: Oral tablets given every 12 hours for 12 weeks
Arm/Group | CF101 1 mg BID | CF101 2 mg BID | CF101 4 mg BID | Placebo
Number analyzed (Participants) | 24 | 17 | 15 | 19
Number of treated patients | 0 | 4 | 1 | 2
Statistical Analysis 1: Comparison: CF101 2 mg BID vs Placebo; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: All adverse events were collected and verbatim terms were coded via MedDRA dictionary
Arm/Group | CF101 1 mg Twice Daily (BID) | CF101 2 mg BID | CF101 4 mg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/17 | 0/15 | 1/19
Other Adverse Events (participants affected / at risk) | 2/24 | 1/17 | 1/15 | 1/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CF101 1 mg Twice Daily (BID) (N=24) | CF101 2 mg BID (N=17) | CF101 4 mg BID (N=15) | Placebo (N=19)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CF101 1 mg Twice Daily (BID) (N=24) | CF101 2 mg BID (N=17) | CF101 4 mg BID (N=15) | Placebo (N=19)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine oxalate (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No